CLINICAL TRIAL: NCT02889978
Title: The Circulating Cell-free Genome Atlas Study
Acronym: CCGA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GRAIL-001
Record Dates: First submitted 2016-08-18; First posted 2016-09-07 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Neoplasms; Cancer
Keywords: Cancer Screening; High-Throughput Nucleotide Sequencing; Deep Sequencing; Circulating cell-free tumor DNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, white blood cells, formalin fixed, paraffin embedded (FFPE) tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cancer arm: Participants with new diagnosis of cancer (multiple tumor types) from which a blood sample and contemporaneous FFPE tumor tissue will be collected.
- Non-cancer arm: Participants with no known diagnosis or past history of cancer from which a blood sample will be collected.

SUMMARY:
GRAIL is using deep sequencing of circulating cell-free nucleic acids (cfNAs) to develop assays to detect cancer early in blood. The purpose of this study is to collect biological samples from participants with a new diagnosis of cancer (blood and tumor tissue) and from participants who do not have a diagnosis of cancer (blood) in order to characterize the population heterogeneity in cancer and non-cancer participants and to develop models for distinguishing cancer from non-cancer.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study with collection of de-identified biospecimens and clinical data from at least 15,000 participants from clinical networks in the United States and Canada. The study will enroll approximately 10,500 cancer participants (CANCER arm) and approximately 4,500 representative participants without a clinical diagnosis of cancer (NON-CANCER arm). Clinical information, demographics, and medical data relevant to cancer status are collected from all participants and their medical record at baseline (time of biospecimen collection), and subsequently from the medical record at intermittent future time points, at least annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria for Non-Cancer Arm Participants:

* Age 20 years or older
* Able to provide a written informed consent

Exclusion Criteria for Non-Cancer Arm Participants:

* Known current or prior diagnosis of cancer except non-melanoma skin cancer
* Oral or IV corticosteroid use in past 14 days prior to blood draw
* Pregnancy (by self-report)
* Current febrile illness
* Acute exacerbation or flare of an inflammatory condition requiring escalation in medical therapy within 14 days prior to blood draw.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant
* Poor health status or unfit to tolerate blood draw

Inclusion Criteria for Cancer Arm Participants:

* Age 20 years or older
* Able to provide a written informed consent

Have either of the following:

A. Confirmed cancer diagnosis (any stage I-IV, as well as carcinoma in situ (CIS) within 90 days prior to or up to 42 days after study blood draw, based upon assessment of a pathological specimen

OR

B. A high suspicion for a cancer diagnosis by clinical and/or radiological assessment, with planned biopsy or surgical resection to establish a definitive diagnosis within 6 weeks (42 days) after study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Known prior diagnosis of cancer except non-melanoma skin cancer
* Currently receiving, or ever received, any of the following therapies to treat their current cancer: surgical management of the cancer beyond that required to establish the cancer diagnosis; local, regional or systemic chemotherapy including chemoembolization; targeted therapy, immunotherapy including cancer vaccines; hormone therapy; or radiation therapy
* Pregnancy (by self-report)
* Current febrile illness
* Acute exacerbation or flare of an inflammatory condition requiring escalation in medical therapy within 14 days prior to blood draw.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant
* Poor health status or unfit to tolerate blood draw

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible study participants will be recruited from participating medical centers in a ratio of 3 non-cancer participants for every 7 cancer participants within each individual research center. Non-cancer subject recruitment will be monitored to achieve demographic characteristics (eg, age, gender, ethnicity, smoking status) reflective of those of the cancer participants.
Sampling Method: Non-Probability Sample
Enrollment: 15254 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
To collect and study clinically-annotated biospecimens, specifically peripheral blood and contemporary tumor tissue when available, to characterize cfNA profiles from deep sequencing and to estimate the population heterogeneity in two arms of the study. | 30 months
To develop and evaluate models for discriminating cancer versus non-cancer and tissue of origin. | 30 months
To evaluate concordance of variants identified in sequencing of tumor tissue and cfNA sequencing results in plasma from the same subject. | 30 months

SECONDARY OUTCOMES:
To explore the relationship between genomic results and clinical outcomes based on collection of longitudinal information (at least annually for up to 5 years) from medical records for all consenting participants. | Year 1, 2, 3, 4, 5
To enable assessment of the performance of an analytically validated clinical laboratory version of the NGS assay (under development) to detect circulating tumor DNA (ctDNA) in plasma. | Year 1, 2, 3, 4, 5

CONTACTS AND LOCATIONS:
Overall Officials: Eric Fung, MD, PhD, Study Director — GRAIL, Inc.
Locations (136):
- United States (135):
  - Southern Cancer Center, PC - Daphne, Daphne, Alabama
  - Southern Cancer Center, P.C. - Mobile Infirmary, Mobile, Alabama
  - Southern Cancer Center, PC - Mobile Airport, Mobile, Alabama
  - Southern Cancer Center, PC - Springhill Medical Center, Mobile, Alabama
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Mercy Fort Smith, Fort Smith, Arkansas
  - Sansum Clinic - 540, Santa Barbara, California
  - Sansum Clinic- 317, Santa Barbara, California
  - Sansum Clinic - Viborg, Solvang, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Center, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Centennial, Colorado
  - Rocky Mountain Cancer Center, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Englewood, Colorado
  - Rocky Mountain Cancer Center, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Hartford HealthCare Cancer Institute at Hartford Hospital, Hartford, Connecticut
  - Hartford New Britain, New Britain, Connecticut
  - UMHC Lennar Foundation - Coral Gables, Coral Gables, Florida
  - UMHC Sylvester- Coral Springs, Coral Springs, Florida
  - University of Miami Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Sylvester at Hollywood, Hollywood, Florida
  - Mayo Clinic - Florida, Jacksonville, Florida
  - University of Miami Sylvester at Kendall, Kendall, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Affiliates - Ocala, Ocala, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - University of Miami Sylvester at Plantation, Plantation, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Maryland Oncology Hematology, P.A., Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Brandywine, Maryland
  - Maryland Oncology Hematology, P.A., Clinton, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Lahey Hospital & Medical Center - Peabody, Peabody, Massachusetts
  - Minnesota Oncology Hematology, P.A. - Main, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, P.A. - Edina, Edina, Minnesota
  - Minnesota Oncology Hematology, P.A. - Woodbury, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Minnesota Oncology Hematology, P.A. - Coon Rapids, Woodbury, Minnesota
  - Mercy Joplin, Joplin, Missouri
  - Mercy Research - Springfield, Springfield, Missouri
  - Memorial Sloan Kettering - Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering, NY - Monmouth, Middletown, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Broome Oncology, LLC, Binghamton, New York
  - New York Oncology Hematology, P.C., Clifton Park, New York
  - Broome Oncology, LLC, Johnson City, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering - Rockville Center, New York, New York
  - Memorial Sloan Kettering, NY - Commack, New York, New York
  - Memorial Sloan Kettering, NY - West Harrison, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Oncology Hematology Care, Inc. - Reading Road, Cincinnati, Ohio
  - Oncology Hematology Care, Inc. - Fairfield, Cincinnati, Ohio
  - Christ Hospital Health Network - The Lindner Center Cancer Research Division, Cincinnati, Ohio
  - Oncology Hematology Care, Inc. - Mercy Health, Cincinnati, Ohio
  - Oncology Hematology Care, Inc. - E. Galbraith, Cincinnati, Ohio
  - Oncology Hematology Care, Inc. - Malsbary, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oncology Hematology Care, Inc. - Five Mile Road, Fairfield, Ohio
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - Northwest Cancer Specialists, P.C. dba Compass Oncology, Portland, Oregon
  - Northwest Cancer Specialists, P.C. dba Compass Oncology, Tualatin, Oregon
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Cancer Center at Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bon Secours Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health - Upstate, Seneca, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Tennessee Oncology Medical Park II, Chattanooga, Tennessee
  - Tennessee Oncology Memorial Plaza, Chattanooga, Tennessee
  - Tennessee Oncology Cleveland Clinic, Cleveland, Tennessee
  - Tennessee Oncology CMC, Crossville, Tennessee
  - Tennessee Oncology Dickson, Dickson, Tennessee
  - Tennessee Oncology Franklin, Franklin, Tennessee
  - Tennessee Oncology Gallatin, Gallatin, Tennessee
  - Tennessee Oncology Summit, Hermitage, Tennessee
  - Tennessee Oncology Lebanon, Lebanon, Tennessee
  - Tennessee Oncology Murfreesboro, Murfreesboro, Tennessee
  - Tennessee Oncology Midtown, Nashville, Tennessee
  - Tennessee Oncology Nashville, Nashville, Tennessee
  - Tennessee Oncology SCCBC, Nashville, Tennessee
  - Tennessee Oncology St. Thomas West, Nashville, Tennessee
  - Tennessee Oncology Skyline, Nashville, Tennessee
  - Tennessee Oncology Southern Hills, Nashville, Tennessee
  - Tennessee Oncology Shelbyville, Shelbyville, Tennessee
  - Tennessee Oncology Stonecrest, Smyrna, Tennessee
  - Texas Oncology - West Texas, Amarillo, Texas
  - Texas Oncology-Bedford, Bedford, Texas
  - TXO - Methodist Dallas Cancer Center, Dallas, Texas
  - Texas Oncology - Dallas Forest Ln, Dallas, Texas
  - Texas Oncology - Presbyterian Cancer Center Dallas, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Fort Worth, Fort Worth, Texas
  - Texas Oncology-Southwest Fort Worth, Fort Worth, Texas
  - Texas Oncology - Grapevine, Grapevine, Texas
  - Texas Oncology Cancer Care and Research Center - Harlingen, Harlingen, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - Mesquite, Mesquite, Texas
  - Texas Oncology-New Braunfels, New Braunfels, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - Plano West, Plano, Texas
  - Texas Oncology - Rockwall, Rockwall, Texas
  - Texas Oncology-San Antonio Downtown, San Antonio, Texas
  - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Texas Oncology-San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology-San Antonio Stone Oak, San Antonio, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Texas Oncology-The Woodlands, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology - Weslaco, Weslaco, Texas
  - Texas Oncology - West Texas, Wichita Falls, Texas
  - Virginia Cancer Specialists, PC, Alexandria, Virginia
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Virginia Cancer Specialists, PC, Woodbridge, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Northwest Cancer Specialists, P.C. dba Compass Oncology, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
- UHN Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mahal BA, Margolis M, Hubbell E, Chen C, Venstrom JM, Abran J, Kartlitz JJ, Wyatt AW, Klein EA. A Targeted Methylation-Based Multicancer Early Detection Blood Test Preferentially Detects High-Grade Prostate Cancer While Minimizing Overdiagnosis of Indolent Disease. JCO Precis Oncol. 2024 Aug;8:e2400269. doi: 10.1200/PO.24.00269. PMID 39208374
- [Derived] Bryce AH, Thiel DD, Seiden MV, Richards D, Luan Y, Coignet M, Zhang Q, Zhang N, Hubbell E, Kurtzman KN, Klein EA. Performance of a Cell-Free DNA-Based Multi-cancer Detection Test in Individuals Presenting With Symptoms Suspicious for Cancers. JCO Precis Oncol. 2023 Jul;7:e2200679. doi: 10.1200/PO.22.00679. PMID 37467458
- [Derived] Tang WHW, Yimer H, Tummala M, Shao S, Chung G, Clement J, Chu BC, Hubbell E, Kurtzman KN, Swanton C, Roberts LR. Performance of a targeted methylation-based multi-cancer early detection test by race and ethnicity. Prev Med. 2023 Feb;167:107384. doi: 10.1016/j.ypmed.2022.107384. Epub 2022 Dec 7. PMID 36495927
- [Derived] Shao SH, Allen B, Clement J, Chung G, Gao J, Hubbell E, Liu MC, Swanton C, Tang WHW, Yimer H, Tummala M. Multi-cancer early detection test sensitivity for cancers with and without current population-level screening options. Tumori. 2023 Jun;109(3):335-341. doi: 10.1177/03008916221133136. Epub 2022 Oct 31. PMID 36316952
- [Derived] Bredno J, Lipson J, Venn O, Aravanis AM, Jamshidi A. Clinical correlates of circulating cell-free DNA tumor fraction. PLoS One. 2021 Aug 25;16(8):e0256436. doi: 10.1371/journal.pone.0256436. eCollection 2021. PMID 34432811
- [Derived] Klein EA, Richards D, Cohn A, Tummala M, Lapham R, Cosgrove D, Chung G, Clement J, Gao J, Hunkapiller N, Jamshidi A, Kurtzman KN, Seiden MV, Swanton C, Liu MC. Clinical validation of a targeted methylation-based multi-cancer early detection test using an independent validation set. Ann Oncol. 2021 Sep;32(9):1167-1177. doi: 10.1016/j.annonc.2021.05.806. Epub 2021 Jun 24. PMID 34176681
- [Derived] Larson MH, Pan W, Kim HJ, Mauntz RE, Stuart SM, Pimentel M, Zhou Y, Knudsgaard P, Demas V, Aravanis AM, Jamshidi A. A comprehensive characterization of the cell-free transcriptome reveals tissue- and subtype-specific biomarkers for cancer detection. Nat Commun. 2021 Apr 21;12(1):2357. doi: 10.1038/s41467-021-22444-1. PMID 33883548
- [Derived] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766